CLINICAL TRIAL: NCT00610103
Title: A Phase 2 Clinical Study of KW-6500 (Apomorphine Hydrochloride) in Patients With Parkinson's Disease
Brief Title: Phase 2 Clinical Study of KW-6500 in Parkinson's Disease Patients With Motor Response Complication on Levodopa Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6500-0702
Record Dates: First submitted 2008-01-22; First posted 2008-02-07 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KW-6500 (Active Comparator): Drug: KW-6500 (apomorphine hydrochloride (USAN))
  Interventions: Drug: apomorphine hydrochloride
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: apomorphine hydrochloride

INTERVENTIONS:
Drug: apomorphine hydrochloride — Apomorphine hydrochloride (started at 1 mg and titrated to a maximum of 6 mg) is subcutaneously administered.
  Other Names: KW-6500

SUMMARY:
The purpose of this study is to evaluate the efficacy of KW-6500 versus placebo when administered as a subcutaneous injection at the individualized maintenance dose level in an OFF state in Parkinson's disease patients with motor response complications on levodopa therapy.

DETAILED DESCRIPTION:
The efficacy of KW-6500 as a subcutaneous injection at the individualized maintenance dose level (1 mg to 6 mg per dose) when used in combination with domperidone (30 mg/day) will be evaluated in comparison with that of placebo in Parkinson's disease patients with motor response complications on levodopa therapy. The maintenance dose level for each subject will be determined using a titration scheme in 1 mg increments.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 years or older at the time of giving informed consent.
* Patients who have idiopathic Parkinson's disease.
* Patients who have been on a stable regimen of levodopa (at least three times daily) plus at least one other antiparkinsonian agent being administered or more frequently for at least 30 days before the preliminary evaluation and who have predictable end-of-dose wearing-off.
* Patients who meet both of the following criteria on the Modified Hoehn and Yahr Scale during the preliminary evaluation and on the day before starting study drug (Day -1).

  * Stage IV or V while in the OFF state
  * Stage II to III while in the ON state
* Patients who have experienced a 30% or more improvement in UPDRS Part 3 score when tested for responsiveness to levodopa during the baseline period.
* Patients who have at least one wearing-off episode per day and a daily average OFF time of at least two hours two days before starting study drug (Day -2) and on Day -1.
* Patients who can understand the OFF state or have a family member who can understand it.
* Patients who have given written informed consent. (Alternatively, the patient's legally acceptable representative may give written consent following the patient's oral consent, if his/her condition makes handwriting difficult.)

Exclusion Criteria:

* Patients with an illness of the cardiac, hematologic, hepatic, renal, pancreatic, metabolic, respiratory, gastrointestinal, endocrinologic, or neurologic system or a tumor that is clinically significant for their participation in the study.
* Patients with orthostatic hypotension.
* Patients with a history of drug allergies.
* Patients with a history of intolerance to morphine or its derivatives, sulfur, sulfur-containing pharmaceutical products, or sulfite.
* Patients with a history of malignant syndrome.
* Patients with a diagnosis of cancer or evidence of continued disease within five years before starting study drug.
* Patients who have been taking domperidone at a dose level of more than 30 mg/day since before the preliminary evaluation.
* Patients who do not test negative in the direct Coombs' test as part of the preliminary evaluation.
* Pregnant or lactating women, women who are planning to have children, women who test positive in the pregnancy test during the preliminary evaluation or on Day -1, or women who cannot adhere to a reliable method of contraception throughout the study.
* Patients who have received MAO inhibitors except selegiline within three months before starting study drug.
* Patients with a current or past history of mental disease or dementia (excluding psychiatric symptoms associated with Parkinson's disease).
* Patients with a Mini-Mental State Examination (MMSE) score of 23 or less on or before Day -1.
* Patients who are taking antipsychotics or dopamine antagonists.
* Patients who are receiving methyldopa, 5-HT3 receptor antagonists, or reserpine.
* Patients who are receiving papaverine.
* Patients who have had a neurosurgical operation for Parkinson's disease.
* Patients who have had transcranial magnetic stimulation (TMS) within six months before starting study drug.
* Patients with a history of drug or alcohol abuse or dependence (DSM-IV criteria) within two years before starting study drug.
* Patients previously treated with apomorphine.
* Patients who have been treated with any other investigational product within four months before starting study drug.
* Patients who, for any reason, are judged by the investigator or subinvestigator to be inappropriate for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The change (response ratio, raw score change, percent score change) in UPDRS (Unified Parkinson's Disease Rating Scale ) Part 3 score at the maintenance dose level | At 20 minutes after administering KW-6500 or placebo

SECONDARY OUTCOMES:
The incidence of adverse events/adverse drug reactions and their nature | 1 week after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (4):
- Japan (4):
  - Tōon, Ehime
  - Tsukuba, Ibaraki
  - Bunkyo-ku, Tokyo
  - Fukuoka